CLINICAL TRIAL: NCT01954420
Title: A Brief Patient-Controlled Intervention for a Symptom Cluster in Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0733; OS11322 (Other: UW Carbone Cancer Center); R01NR013468-01A1 (NIH); 2013-0733 (Other: Institutional Review Board); A549000 (Other: UW Madison); NUR\RESEARCH\NURSNG RES (Other: UW Madison); NCI-2013-02325 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2017-02

CONDITIONS: Pain; Fatigue; Sleep Disturbance; Cancer
Keywords: Pain; Fatigue; Sleep; Cancer; Relaxation; Distraction; Symptoms
MeSH Terms: conditions — Pain; Fatigue; Parasomnias; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Control (Other): Standard care + cancer education
  Participants receive a single session with a research nurse to discuss the importance of understanding cancer and cancer treatment strategies, and to introduce educational recordings available on an MP3 player. The educational recordings provide a selection of publicly available American Cancer Society patient information materials addressing topics related to cancer and cancer treatment strategies. Participants are asked to listen to at least one recording per day, or more frequently as desired.
  Interventions: Other: Attention Control
- Cognitive-Behavioral Intervention (Experimental): Standard care + Patient-Controlled Cognitive Behavioral Intervention
  Participants will receive a single training session with a research nurse including: 1) Information about the causes of cancer-related pain, fatigue, and sleep disturbance. 2) An explanation of how cognitive-behavioral interventions may affect symptoms. 3) Review of the specific cognitive-behavioral strategies provided on the MP3 player. 4) Individualized recommendations for using the cognitive-behavioral strategies. The nurse interventionist and patient will develop a written plan for practicing the strategies with recommendations to use a strategy at least once a day, or more frequently as needed.
  Interventions: Behavioral: Cognitive-Behavioral Intervention

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention — Standard care + Selection of 12 recorded imagery- and non imagery-based cognitive-behavioral coping strategies provided on an MP3 player.
  Arms: Cognitive-Behavioral Intervention
Other: Attention Control — Standard care + Cancer education
  Arms: Attention Control

SUMMARY:
The purpose of the research is to test the efficacy of a patient-controlled cognitive-behavioral intervention for pain, fatigue, and sleep disturbance during cancer treatment, and to evaluate moderators and mediators of intervention effects. The intervention uses guided imagery, relaxation exercises, and nature sound recordings, self-administered via an MP3 player. The study will determine (1) if the intervention helps to control symptoms during chemotherapy, (2) if personal and clinical characteristics influence how well the intervention works, and (3) if the cognitive-behavioral strategies reduce markers of stress and inflammation found in blood and saliva.

DETAILED DESCRIPTION:
Co-occuring pain, fatigue, and sleep disturbance is a common symptom cluster among patients with advanced cancer, diminishing functional status and quality of life. Cognitive-behavioral (CB) strategies (e.g., relaxation, distraction, and imagery) are effective treatments for each of these symptoms, and provide a logical choice in managing all three co-occurring symptoms. CB strategies are thought to work psychologically by reducing anxiety and stress, improving expectations for symptom outcomes, and enhancing perceptions of personal control. Recent research also suggests a physiologic pathway, in which CB strategies attenuate dysregulation in stress hormones and reduce proinflammatory cytokines that contribute to symptom exacerbation. CB strategies are not equally effective for all patients, with differences based on individual preferences and skills and concurrent symptoms. Thus, training in a single strategy is not sufficient. Our previous work demonstrates feasibility and initial efficacy of a patient-controlled cognitive-behavioral (PC-CB) intervention in which patients receive information about their symptoms and rationale for CB strategies, then self-administer their selection of various relaxation, distraction, and imagery strategies via MP3 player, using the CB strategies at whatever time and place they are needed. This brief intervention was designed to be mindful of the high symptom burden, unpredictable treatment course, and often short life expectancy of persons with advanced cancer. The purpose of this study is to test efficacy of the PC-CB intervention in a randomized controlled trial and to test moderators and mediators of intervention effects. The specific aims are (1) to test efficacy of the PC-CB intervention on severity, distress, and interference with daily life from the pain, fatigue, sleep disturbance symptom cluster, (2) to test proposed moderators (imaging ability, concurrent symptoms) of PC-CB intervention effects, (3) to test psychological mediators (anxiety, stress, outcome expectancy, perceived control) of PC-CB intervention effects, and (4) to explore two types of physiological mediators (neuroendocrine stress hormones and indices of inflammation) of PC-CB intervention effects. A sample of 198 adults receiving chemotherapy for advanced breast, lung, colorectal, prostate, gynecologic or other solid tumor cancers and experiencing pain, fatigue, and sleep disturbance will be recruited. Patients randomized to the PC-CB intervention will receive a brief training session and instructions to use the recorded CB strategies during 9-weeks of cancer treatment. Patients randomized to attention control will receive instructions to use cancer educational recordings over the same period. Measures of symptom severity and distress, symptom interference with daily life, and proposed psychological and physiologic mediating variables will be completed at baseline and the 3-week (primary) time point. Symptom outcome measures will be repeated at 6- and 9-week (secondary) time points to evaluate longer term treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Have a diagnosis of advanced (metastatic or recurrent) lung, breast, colorectal, prostate, gynecologic or other solid tumor cancer.
* Be receiving outpatient chemotherapy.
* Report all three symptoms (pain, fatigue, and sleep disturbance) as present in the past week with worst severity rating ≥ 3 (0-10 scale) for at least two of the three symptoms -

Exclusion Criteria:

* Pain that is post-operative (< 3 months since surgery) or severe neuropathic pain.
* Hospitalized for psychiatric reasons within the past 3 months.
* Unable to read, write, or understand English, or otherwise unable to complete study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Symptom Cluster Severity | 3-weeks
Symptom Cluster Distress | 3-weeks
Symptom Cluster Interference with Daily Life | 3-weeks

SECONDARY OUTCOMES:
Symptom Cluster Severity | 6- and 9-weeks
Symptom Cluster Distress | 6- and 9-weeks
Symptom Cluster Interference with Daily Life | 6- and 9-weeks

OTHER OUTCOMES:
Quality of Life | 3-, 6-, 9-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Kwekkeboom, PhD., RN, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - SwedishAmerican Regional Cancer Center, Rockford, Illinois
  - Mercy Health System, Janesville, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/